CLINICAL TRIAL: NCT02834936
Title: A Phase 2 Clinica Study: Efficacy and Safety of Pyrotinib in Patients of Advanced Non-Small Cell Lung Cancer With HER2 Mutation
Brief Title: A Clinica Study of Pyrotinib in Patients of Advanced Non-Small Cell Lung Cancer With HER2 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-Ⅱ-NSCLC
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pyrotinib treatment (Experimental)
  Interventions: Drug: pyrotinib

INTERVENTIONS:
Drug: pyrotinib
  Other Names: BLTN

SUMMARY:
This study is designed to evaluate the efficacy and safety of Pyrotinib in patients of advanced pre-treated Non-small cell lung cancer With HER2 Mutation.

To observe objective response rate (ORR) of pyrotinib in NSCLC With HER2 Mutation. To observe Progression free survival (PFS). To assess the overall survival (OS).

A secondary aim is to obtain safety information.

To explore the relationship between biomarkers and the toxicity/efficacy of Pyrotinib.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status of 0 to 1.
2. Life expectancy of more than 3 months.
3. At least one measurable lesion exists.(RECIST 1.1).
4. Histologically or cytologic confirmed Non-small cell lung cancer, Phase IIIB or IV according to IASLC 2009.
5. Failed prior therapies.(RECIST 1.1).
6. Confirmed HER2 mutation by Central Laboratory。
7. More than one prior Platinum based chemotherapy for advanced and/or metastatic, or recurrent NSCLC in neoadjuvant or adjuvant chemotherapy.
8. Required laboratory values including following parameters:

   ANC: ≥ 1.5 x 10^9/L; Platelet count: ≥ 90 x 10^9/L; Hemoglobin: ≥ 90 g/L; Total bilirubin: ≤ 1.5 x upper limit of normal (ULN); ALT and AST: ≤2 x ULN or ALT and AST: ≤5x ULN for patients with liver metastasis; BUN and Cr: ≤1.5 x ULN； creatine clearance rate: ≥ 50 mL/min; LVEF: ≥ 50%; QTcF: < 470 ms for female and < 450 ms for male.
9. Signed informed consent

Exclusion Criteria:

1. Previous therapy with other HER2 inhibitors.
2. History of severe hypersensitivity reactions to the excipients of the trial drugs.
3. Have clinically significant cavity effusion,such as pleural effusion、 pericardial effusion or ascites and require clinical intervention
4. Active brain metastases
5. Other malignancy within the past (including primary brain tumor or Leptomeningeal tumor), other than basal cell skin cancer or carcinoma in situ of the cervix
6. Persistence of clinically relevant therapy related toxicities from previous therapy (greater than Common Terminology Criteria for Adverse Event(CTCAE) 4.0 grade 1)
7. Treatment with surgery, chemotherapy, radiotherapy or other target therapy within the past 4 weeks before start of therapy
8. Uncontrolled hypertensin,diabetes.
9. unstable angina, history of myocardial infarction in the past 6 months, congestive heart failure>NYHA II, serious cardiac arrhythmia
10. Active infection
11. Variety of factors that affect the oral medication (such as unable to swallow, chronic diarrhea, bowel obstruction and other gastrointestinal disorders or abnormalities
12. History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
13. Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
14. Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
15. Known history of neurological or psychiatric disease, including epilepsy or dementia.
16. Treatment in another clinical trial within the past 4 weeks before start of therapy
17. Any of the other conditions of which researchers believe that the patient is not fit to take part in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | tumor assessment every 6-9 weeks after the initiation of pyrotinib, up to 24 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months
Incidence and Intensity of Adverse Events | From signing informed consent document until 28 days after the last drug administration
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - HR-BLTN-II-NSCLC Investigational Site, Beijing
  - HR-BLTN-II-NSCLC Investigational Site, Changsha
  - HR-BLTN-II-NSCLC Investigational Site, Guangzhou
  - HR-BLTN-II-NSCLC Investigational Site, Hangzhou
  - HR-BLTN-II-NSCLC Investigational Site, Harbin
  - HR-BLTN-II-NSCLC Investigational Site, Nanjing
  - HR-BLTN-II-NSCLC Investigational Site, Shanghai
  - HR-BLTN-II-NSCLC Investigational Site, Suzhou
  - HR-BLTN-II-NSCLC Investigational Site, Wuhan
  - HR-BLTN-II-NSCLC Investigational Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided
The plan havn't been decided

REFERENCES:
- [Derived] Mao S, Yang S, Liu X, Li X, Wang Q, Zhang Y, Chen J, Wang Y, Gao G, Wu F, Jiang T, Zhang J, Yang Y, Lin X, Zhu X, Zhou C, Ren S. Molecular correlation of response to pyrotinib in advanced NSCLC with HER2 mutation: biomarker analysis from two phase II trials. Exp Hematol Oncol. 2023 Jun 9;12(1):53. doi: 10.1186/s40164-023-00417-y. PMID 37296463
- [Derived] Zhou C, Li X, Wang Q, Gao G, Zhang Y, Chen J, Shu Y, Hu Y, Fan Y, Fang J, Chen G, Zhao J, He J, Wu F, Zou J, Zhu X, Lin X. Pyrotinib in HER2-Mutant Advanced Lung Adenocarcinoma After Platinum-Based Chemotherapy: A Multicenter, Open-Label, Single-Arm, Phase II Study. J Clin Oncol. 2020 Aug 20;38(24):2753-2761. doi: 10.1200/JCO.20.00297. Epub 2020 Jul 2. PMID 32614698